CLINICAL TRIAL: NCT02547324
Title: Slump Sitting X-ray of the Lumbar Spine Is Better Than Conventional Flexion
Brief Title: Slump Sitting X-ray of the Lumbar Spine Is Better Than Conventional Flexion View
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study results were too significant
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Orthosurgery, Dr. Hey Hwee Weng Dennis, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2013/00141
Record Dates: First submitted 2015-08-20; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Low Back Pain; Spondylolisthesis
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slump sitting (Experimental): Slump sitting flexion of lumbar spine
  Interventions: Radiation: Slump sitting
- Forward bending (Active Comparator): Forward erect bending of lumbar spine
  Interventions: Radiation: Forward bending

INTERVENTIONS:
Radiation: Slump sitting — Patients are asked to sit slumped on the chair as much as possible without leaning forwards, and place you hands below your thighs.
  Arms: Slump sitting
Radiation: Forward bending — Patients are asked to stand with both feet placed together, hands behind their heads, and bend forward in this position as much as possible without falling
  Arms: Forward bending

SUMMARY:
This is a prospective, single-blinded, randomized-controlled study comparing a new method (slump-sitting) with the conventional method (forward erect bending) of performing lumbar spine flexion X-rays.

DETAILED DESCRIPTION:
Power calculation was performed based on preliminary pilot results using a clinically set difference of 10 degrees (SD 15 degrees) change in mean global lumbar spine flexion between sitting and standing postures. An estimated sample population of 100 patients was deemed necessary for this study to fulfill a statistical power of 90% and a two-sided 5% significance level.

Block randomization of every 4 subjects was performed at the beginning of the study to ensure equal numbers of subjects in both study arms for comparison and these results were concealed in envelopes.

During the clinical consult, history taking was performed as per a usual clinic visit. Specific patient's details including age, occupation, presence and severity of back pain, presence and severity of leg pain, and neurological symptoms were documented. Physical examination was performed accordingly and parameters such as clinical range of motion of the lumbar spine, neurological signs and provocative tests were recorded for later analysis.

For the flexion radiographs, both the new and conventional methods were performed on each patient. These pictures were made into charts and visually displayed. They serve as instructional manuals for patients during the radioimaging process, which are again reinforced with verbal instructions from the on-duty radiographers.

Both images were done with the X-ray beam projected from the patients's left and at a distance of 100cm from the patient. The central beam was directed at the estimated centre of L3, with T11 vertebral body and mid-body of the sacrum serving as superior and inferior limits respectively. A single extension view of the lumbar spine was also performed after these flexion views. All radiographs were stored on Digital Imaging and Communications in Medicine (DICOM) format and viewed with Centricity Enterprise Web V3.0 (8.0.1400.128) for assessment.

Measurements were done by 2 independent reviewers and an average of their readings was recorded. Both reviewers were blinded to the method in which flexion X-rays was taken.

Interim data analysis is planned at 30th patient and the 60th patient. During this time point, the primary objective which look at mean global lumbar spine flexion between sitting and standing postures is assessed.

All collected data and measurements were tabulated using Microsoft Excel 2011(Version 14.0 (32-bit)) and analyzed using International Business Machines (IBM) Statistical Package for the Social Sciences (SPSS Version 23.0).

For the main analysis of both global and segmental lumbar flexion, as well as the measured displacements obtained between the two flexion methods, paired t-test was employed.

There is no requirement to follow up the patients in this study. The whole study is to be completed within 1 year of recruitment

ELIGIBILITY:
Inclusion Criteria:

* Patients above 45 years of age;
* With mechanical low back pain,
* With spondylolisthesis
* Physically able to position themselves correctly for both methods of X-rays

Exclusion Criteria:

* Previous spinal interventions
* Suspected findings for spinal malignancies, spinal trauma, and inflammatory spinal diseases
* Pregnant women

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Global lumbar spine flexion range of motion | Day 1 (no follow-up, outcome assessed immediately)
  Change in mean global lumbar spine flexion between sitting and standing postures

SECONDARY OUTCOMES:
Segmental lumbar spine flexion range of motion | Day 1 (no follow-up, outcome assessed immediately)
  Change in segmental global lumbar spine flexion between sitting and standing postures
Segmental translational changes during lumbar spine flexion | Day 1 (no follow-up, outcome assessed immediately)
  Percentage translation at each segmental lumbar spine levels

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Kit Wong, MBBS, Study Chair — National University Health System